CLINICAL TRIAL: NCT02526368
Title: A Pilot Study of Magnetic Resonance (MR) Imaging with Hyperpolarized Pyruvate (13C) to Detect High Grade Localized Prostate Cancer
Brief Title: Pilot Study of (MR) Imaging with Pyruvate (13C) to Detect High Grade Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ivan de Kouchkovsky, MD (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor-Investigator, Ivan de Kouchkovsky, MD, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15557; NCI-2015-02008 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA211150 (NIH); U01EB026412 (NIH)
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Localized Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Pre-surgical Prostate Cancer patients (Experimental): Participants will receive an infusion of hyperpolarized 13C-pyruvate alone or co-hyperpolarized 13C pyruvate with hyperpolarized 13C, 15N urea injection prior to metabolic/perfusion high spatial resolution MRI/1H MRSI staging exam (PROSE) with endorectal coil using both a phased-array abdominal coil and an endorectal coil will be performed within 12 weeks of subsequent non-investigational radical prostatectomy.
- Cohort B: Post-HIFU Participants (Experimental): Participants will receive an infusion of hyperpolarized 13C-pyruvate alone or co-hyperpolarized 13C pyruvate with hyperpolarized 13C, 15N urea injection prior to metabolic/perfusion high spatial resolution MRI/1H MRSI staging exam (PROSE) with endorectal coil using both a phased-array abdominal coil and an endorectal coil will be performed for participants with planned post-HIFU surveillance systematic and MR-targeted non-investigational biopsies

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Given IV
  Other Names: Hyperpolarized Pyruvate (13C)
Drug: Hyperpolarized 13C,15N2-urea — Given IV
  Other Names: Urea C-13; C13 Urea
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: MRSI; MRS; 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; MRS Imaging

SUMMARY:
This pilot clinical trial studies how well magnetic resonance spectroscopic imaging (MRSI) with hyperpolarized carbon 13 (13C) pyruvate alone or in combination with 13C 15N2 Urea works in finding prostate cancer that exhibits poorly differentiated or undifferentiated cells (high-grade) and that is restricted to the site of origin, without evidence of spread (localized) in patients undergoing radical prostatectomy. Diagnostic procedures, such as MRSI with hyperpolarized carbon (13C) pyruvate, may aid in the diagnosis of prostate cancer and in discriminating high-grade from low-grade prostate cancer and benign adjacent prostate tissue

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the association between hyperpolarized (HP) pyruvate-to-lactate conversion (kPL) and HP urea perfusion with histologic grade of prostate cancer, including benign prostate tissue, low grade disease (primary Gleason score < 4), and high grade (primary Gleason score >= 4) prostate cancer (Cohort A).

II. To investigate the association between HP pyruvate-to-lactate conversion (kPL) and HP urea perfusion with in-field clinically significant (Gleason score >3+3) recurrent/residual prostate cancer following non-investigational High-Intensity Focused Ultrasound (HIFU) focal therapy (Cohort B)

SECONDARY OBJECTIVES:

I. Safety.

II. To determine the optimal cut-off value of peak lactate to pyruvate ratio (lac/pyr), lac/pyr area under the curve (AUC), 13C pyruvate to lactate (kPL) rate, urea AUC, and urea transfer constant (ktrans) on magnetic resonance imaging (MRI) that accurately detects primary Gleason 4 component cancer (Cohort A).

III. To determine the optimal cut-off value of peak lac/pyr, lac/pyr AUC, kPL Urea AUC, Urea ktrans and kPL-urea product (kUP) on MRI that accurately detects in-field clinically significant (ie. Gleason score >3+3) recurrent/residual prostate cancer (Cohort B only).

IV. To determine the reproducibility of peak lac/pyr, lac/pyr AUC and kPL, urea AUC and urea transfer constant (ktrans) with same-day repeated dose studies. with same-day repeated dose studies.

V. To compare peak lac/pyr, lac/pyr AUC and kPL, urea AUC, urea transfer constant (ktrans) on MRI with Prostate Imaging-Reporting and Data System (PI-RADS) assessment of multiparametric MRI in predicting regions of cancer versus benign tissue.

EXPLORATORY OBJECTIVES:

I. To correlate histologic markers, including lactate dehydrogenase A (LDHA) expression and activity level, along with Ki-67, MYC, and MCT 1 and 4 expression, with peak intra-tumoral lac/pyr ratio, lactate AUC, and kPL detected using anatomically aligned magnetic resonance (MR) cross-sectional images of the prostate gland.

II. To test for an association between mean intra-tumoral lac/pyr signal and lactate AUC, kPL, urea AUC, and urea transfer constant (ktrans) with adverse clinical and pathologic characteristics including extracapsular extension, positive nodal involvement, and failure to achieve undetectable prostate specific antigen (PSA) nadir following prostatectomy.

OUTLINE:

Participants receive either hyperpolarized carbon pyruvate (13C) or co-polarized 13C pyruvate and 13C, 15N2urea intravenously (IV) and undergo MRSI within 12 weeks of undergoing non-investigational radical prostatectomy (cohort A) or non-investigational systematic and MR-targeted biopsies (cohort B). Participants may receive optional second hyperpolarized 13C injection and dynamic 13C MRI scan performed within 15 to 60 minutes following completion of first scan.

After completion of study, participants are followed up at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the prostate. Biopsy may be performed outside of University of California, San Francisco (UCSF), if detailed results of sextant biopsy are available. For Cohort A only, a minimum of 20 participants out of a planned enrollment of 50 patients must have high-risk disease as defined by primary Gleason score of 4 or 5 on prior prostate biopsy.
* Cohort A only: Planned radical prostatectomy at UCSF within 12 weeks following protocol MRI/MRSI.
* Cohort B only: HIFU focal therapy completed within 18 months of protocol MRI/MRSI, and planned systematic and MR-guided biopsy at UCSF within 12 weeks following protocol MRI/MRSI.
* The participant is able and willing to comply with study procedures and provide signed and dated informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1500 cells/microliter (uL)
* Hemoglobin >= 9.0 mg/dL
* Platelets >= 75,000 cells/uL
* Estimated creatinine clearance >= 50 mL/min (by the Cockcroft Gault equation)
* Bilirubin < 1.5 x upper limit of normal (ULN) (unless Gilbert's is suspected)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x ULN

Exclusion Criteria:

* Participants who because of age less than 18 years old, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
* Participants unwilling or unable to undergo MR imaging, including patients with contraindications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
* Participants who cannot tolerate or have contra-indications to endorectal coil insertion; for example, participants with a prior abdominoperineal resection of the rectum or latex allergy.
* Patients with contra-indications to injection of gadolinium contrast; for example patients with prior documented allergy or those with inadequate renal function.
* Metallic hip implant or any other metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging.
* Cryosurgery, surgery for prostate cancer, prostatic or pelvic radiotherapy prior to study enrollment. For Cohort B, HIFU focal therapy is allowed. No limit on number of prior prostate biopsies; prior transurethral prostatic resection (TURP) is not allowed.
* Current or prior androgen deprivation therapy. For Cohort A, a history of use of a 5-alpha reductase inhibitor is allowed, provided it was discontinued at least one month prior to study entry. For cohort B, a history of use of 5-α reductase inhibitor is allowed, provided it is discontinued at least 14 days to protocol MRI/MRSI.
* Poorly controlled hypertension, with blood pressure at study entry > 160/100; the addition of anti-hypertensives to control blood pressure is allowed for eligibility determination.
* Congestive heart failure or New York Heart Association (NYHA) status >= 2.
* A history of clinically significant electrocardiography (EKG) abnormalities, including QT prolongation, a family history of prolonged QT interval syndrome, or myocardial infarction (MI) within 6 months of study entry; patients with rate-controlled atrial fibrillation/flutter will be allowed on study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-03-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean peak intra-tumoral lactate/pyruvate (lac/pyr) ratio by pathological grade (Cohort A) | Baseline, 1 day
  Means and standard deviations for lactate area under curve will be calculated by pathologic grade (benign, low grade (primary Gleason score <4) and high grade (primary Gleason score >4)).
Mean peak intra-tumoral lactate/pyruvate (lac/pyr) ratio (Cohort B) | Baseline, 1 day
  Means and standard deviations for lactate area under curve will be calculated for those with in-field recurrent/residual clinically significant prostate cancer.
Mean lactate area under curve (AUC) by pathological grade (Cohort A) | Baseline, 1 day
  Means and standard deviations for lactate area under curve will be calculated by pathologic grade (benign, low grade (primary Gleason score <4) and high grade (primary Gleason score >4)). A One-way ANOVA model will be used to compare lactate area under curve by pathologic grade (benign, low grade (primary Gleason score <4) and high grade (primary Gleason score >4)).
Mean lactate area under curve (AUC) (Cohort B) | Baseline, 1 day
  Means and standard deviations for lactate area under curve will be calculated for those with in-field recurrent/residual clinically significant prostate cancer.
Mean peak conversion of HP 13C pyruvate to lactate (kPL) by pathological grade (Cohort A) | Baseline, 1 day
  Means and standard deviations for kPL will be calculated by pathologic grade (benign, low grade (primary Gleason score <4) and high grade (primary Gleason score >4)).
Mean peak conversion of HP 13C pyruvate to lactate (kPL) (Cohort B) | Baseline, 1 day
  Means and standard deviations for kPL will be calculated for those with in-field recurrent/residual clinically significant prostate cancer.
Mean Urea AUC by pathological grade (Cohort A) | Baseline, 1 day
  Means and standard deviations for Urea AUC will be calculated by pathologic grade (benign, low grade (primary Gleason score <4) and high grade (primary Gleason score >4)).
Mean Urea AUC (Cohort B) | Baseline, 1 day
  Means and standard deviations for Urea AUC will be calculated for those with in-field recurrent/residual clinically significant prostate cancer.
Mean urea transfer constant (Ktrans) by pathological grade (Cohort A) | Baseline, 1 day
  Means and standard deviations for Ktrans will be calculated by pathologic grade (benign, low grade (primary Gleason score <4) and high grade (primary Gleason score >4)).
Mean urea transfer constant (Ktrans) (Cohort B) | Baseline, 1 day
  Means and standard deviations for Ktrans will be calculated for those with in-field recurrent/residual clinically significant prostate cancer.

SECONDARY OUTCOMES:
Optimal cut-off value of peak lactate to pyruvate ratio (lac/pyr) (Cohort A) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of peak lac/pyr AUC on MRI that accurately detect primary Gleason 4 prostate cancer.
Optimal cut-off value of peak lactate to pyruvate ratio (lac/pyr) (Cohort B) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of peak lac/pyr AUC on MRI that accurately detects in-field clinically significant (i.e. Gleason score >3+3) recurrent/residual prostate cancer.
Optimal cut-off value of lac/pyr area under the curve (AUC) (Cohort A) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of peak lac/pyr AUC values on MRI that accurately detect primary Gleason 4 prostate cancer
Optimal cut-off value of lac/pyr area under the curve (AUC) (Cohort B) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of peak lac/pyr AUC values on MRI that accurately detects in-field clinically significant (ie. Gleason score >3+3) recurrent/residual prostate cancer
Optimal cut-off value of 13C pyruvate to lactate (kPL) rate (Cohort A) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of kPL on MRI that accurately detect primary Gleason 4 prostate cancer.
Optimal cut-off value of 13C pyruvate to lactate (kPL) rate (Cohort B) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of kPL on MRI that accurately detects in-field clinically significant (ie. Gleason score >3+3) recurrent/residual prostate cancer
Optimal cut-off value of urea AUC (Cohort A) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of urea AUC on MRI that accurately detect primary Gleason 4 prostate cancer.
Optimal cut-off value of urea AUC (Cohort B) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of urea AUC on MRI that accurately detects in-field clinically significant (ie. Gleason score >3+3) recurrent/residual prostate cancer
Optimal cut-off value of urea transfer constant (ktrans) (Cohort A) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of urea ktrans on MRI that accurately detect primary Gleason 4 prostate cancer.
Optimal cut-off value of urea transfer constant (ktrans) (Cohort B) | Baseline, 1 day
  Receiver-operative-curve analyses will be performed to determine the optimal cut-point of urea ktrans on MRI that accurately detects in-field clinically significant (ie. Gleason score >3+3) recurrent/residual prostate cancer
Proportion of participants with Treatment-Related Adverse Events | Baseline, 1 day
  Assessment of the occurrence of clinically significant changes in safety variables from baseline. Safety endpoints include monitoring for the occurrence of treatment-emergent AEs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology (Toxicity) Criteria for Adverse Events (CTCAE) version 4.0.
Compare lactate/pyruvate area under curve (AUC) with Prostate Imaging Reporting and Data System (PI-RADS) | Baseline, 1 day
  To compare lactate/pyruvate AUC on MRI with PI-RADS assessment of multiparametric MRI in predicting regions of cancer versus benign tissue. Radiologists use the PI-RADS to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious).
Compare peak lactate/pyruvate with PI-RADS | Baseline, 1 day
  To compare peak lactate/pyruvate on MRI with PI-RADS assessment of multiparametric MRI in predicting regions of cancer versus benign tissue. Radiologists use the PI-RADS to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious).
Compare pyruvate to lactate (kPL) with PI-RADS | Baseline, 1 day
  To compare peak pyruvate to lactate (kPL) on MRI with PI-RADS assessment of multiparametric MRI in predicting regions of cancer versus benign tissue. Radiologists use the PI-RADS to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious).
Compare urea AUC with PI-RADS | Baseline, 1 day
  To compare urea AUC on MRI with PI-RADS assessment of multiparametric MRI in predicting regions of cancer versus benign tissue. Radiologists use the PI-RADS to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious).
Compare urea transfer constant (Ktrans) with PI-RADS | Baseline, 1 day
  To compare urea ktrans on MRI with PI-RADS assessment of multiparametric MRI in predicting regions of cancer versus benign tissue. Radiologists use the PI-RADS to report how likely it is that a suspicious area is a clinically significant cancer. PI-RADS scores range from 1 (most likely not cancer) to 5 (very suspicious).
Mean difference in Intra-patient peak lac/pyr | Baseline, 1 day
  Intra-patient reproducibility of peak lac/pyr for patients who undergo repeated dose imaging studies, as descriptively reported using summary statistics.
Mean difference in Intra-patient lac/pyr AUC | Baseline, 1 day
  Intra-patient reproducibility of lac/pyr AUC for patients who undergo repeated dose imaging studies, as descriptively reported using summary statistics.
Mean difference in Intra-patient kPL | Baseline, 1 day
  Intra-patient reproducibility of kPL for patients who undergo repeated dose imaging studies, as descriptively reported using summary statistics.
Mean difference in Intra-patient Urea AUC | Baseline, 1 day
  Intra-patient reproducibility of Urea AUC for patients who undergo repeated dose imaging studies, as descriptively reported using summary statistics.
Mean difference in Intra-patient Urea ktrans | Baseline, 1 day
  Intra-patient reproducibility of Urea ktrans for patients who undergo repeated dose imaging studies, as descriptively reported using summary statistics

CONTACTS AND LOCATIONS:
Overall Officials: Ivan de Kouchkovsky, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No